CLINICAL TRIAL: NCT01157351
Title: A Fifteen-month, Prospective, Randomized, Active-controlled, Open-label, Flexible Dose Study of Paliperidone Palmitate Compared With Oral Antipsychotic Treatment in Delaying Time to Treatment Failure in Adults With Schizophrenia Who Have Been Incarcerated
Brief Title: 15 Month Study for Adults Who Have Been Diagnosed With Schizophrenia and Incarcerated
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR015625; R092670SCH3006 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2010-05-03; First posted 2010-07-07 (Estimated); Results first posted 2014-12-04 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Risperidone; Risperdal; Paliperidone palmitate; Aripiprazole; Haloperidol; Olanzapine; Paliperidone; Perphenazine; Quetiapine
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate; Risperidone; Perphenazine; Aripiprazole; Quetiapine Fumarate; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- 001 (Experimental): paliperidone palmitate 78 117 156 or 234 mg monthly injection for 15 months
  Interventions: Drug: paliperidone palmitate
- 002 (Active Comparator): aripiprazole flexible dosing as prescribed by the study doctor for 15 months
  Interventions: Drug: aripiprazole
- 003 (Active Comparator): haloperidole flexible dosing as prescribed by the study doctor for 15 months
  Interventions: Drug: haloperidole
- 004 (Active Comparator): olanzapine flexible dosing as prescribed by the study doctor for 15 months
  Interventions: Drug: olanzapine
- 005 (Active Comparator): paliperidone flexible dosing as prescribed by the study doctor for 15 months
  Interventions: Drug: paliperidone
- 006 (Active Comparator): perphenazine flexible dosing as prescribed by the study doctor for 15 months
  Interventions: Drug: perphenazine
- 007 (Active Comparator): quetiapine flexible dosing as prescribed by the study doctor for 15 months
  Interventions: Drug: quetiapine
- 008 (Active Comparator): risperidone flexible dosing as prescribed by the study doctor for 15 months
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: paliperidone — flexible dosing as prescribed by the study doctor for 15 months
  Arms: 005
Drug: risperidone — flexible dosing as prescribed by the study doctor for 15 months
  Arms: 008
Drug: haloperidole — flexible dosing as prescribed by the study doctor for 15 months
  Arms: 003
Drug: perphenazine — flexible dosing as prescribed by the study doctor for 15 months
  Arms: 006
Drug: aripiprazole — flexible dosing as prescribed by the study doctor for 15 months
  Arms: 002
Drug: quetiapine — flexible dosing as prescribed by the study doctor for 15 months
  Arms: 007
Drug: paliperidone palmitate — 78, 117, 156, or 234 mg monthly injection for 15 months
  Arms: 001
Drug: olanzapine — flexible dosing as prescribed by the study doctor for 15 months
  Arms: 004

SUMMARY:
The study will assess the use of paliperidone palmitate compared with oral antipsychotic treatment in delaying time to a protocol-defined treatment failure over 15 months, in patients diagnosed with schizophrenia who have been incarcerated.

DETAILED DESCRIPTION:
The primary objective of this study is to compare the efficacy of paliperidone palmitate with oral antipsychotic treatment in delaying time to a protocol-defined treatment failure over 15 months, in patients diagnosed with schizophrenia who have been incarcerated. Protocol-defined treatment failure is defined as arrest, psychiatric hospitalization, increase in psychiatric services to prevent imminent hospitalization, discontinuation of antipsychotic treatment due to inadequate efficacy, treatment supplementation with another antipsychotic due to inadequate efficacy, discontinuation of antipsychotic treatment due to safety or tolerability or completed suicide. Protocol was amended on March 15, 2011 to reflect changes in the inclusion/exclusion criteria as well as the study objectives. Patients will receive either paliperidone palmitate 78, 117, 156, or 234 mg monthly by injection for fifteen months OR oral aripiprazole, haloperidol, olanzapine, paliperidone, perphenazine, quetiapine, and risperidone at doses selected by the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to understand and sign the informed consent form approved by the Institutional Review Board (IRB)
* Must successfully answer all the questions on the Informed Consent quiz indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study
* Have a current diagnosis of schizophrenia
* Taking no more than 1 oral antipsychotic on the day before randomization
* Have been placed into custody at least twice with one of them leading to incarceration within the 24 months previous to study start, with the last release occurring within the 90 days before the first day of screening
* in the opinion of the investigator, may benefit from a change in their prior antipsychotic treatment
* Have available a designated individual (eg, family member, case manager, significant other, probation/parole officer) who has knowledge of the patient and is generally aware of the patient's daily activities, and who agrees to let the study site personnel know of changes in the patients circumstances when the patient is not able to provide this information, ie, arrests, protocol-defined hospitalizations, emergency room visits, becoming homeless, etc.
* Have either an address or phone number where they can be reached, or be accessible to the designated individual
* Must agree to receive regular injections for 15 months if randomly assigned to the paliperidone palmitate treatment group, or continue with oral study medication treatment for 15 months if randomly assigned to the oral antipsychotic treatment group
* Women must be postmenopausal (for at least 2 years), surgically sterile (hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), abstinent, or if sexually active, be practicing a highly effective method of birth control

Exclusion Criteria:

* Allergies, hypersensitivity (anaphylaxis-type reaction), or intolerance to risperidone or paliperidone
* Actively abusing intravenous drugs within the past 3 months or have an opiate dependence disorder
* Have a positive urine drug screen test for barbiturates, cocaine, amphetamines, or opiates at screening
* Women who are pregnant or breast-feeding, or planning to become pregnant
* Have received injectable antipsychotic treatment within 2 injection cycles prior to screening
* Received treatment with clozapine within 3 months of screening
* Are at a high risk of violence in the next 15 months, in the opinion of the investigator
* who have a history of sex offenses including felony sex offenses, child molestation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2010-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (56):
- United States (55):
  - Bullhead City, Arizona
  - Tuscon, Arizona
  - Little Rock, Arkansas
  - Anaheim, California
  - Escondido, California
  - Glendale, California
  - Imperial, California
  - Long Beach, California
  - National City, California
  - Oakland, California
  - Oceanside, California
  - Pico Rivera, California
  - Riverside, California
  - San Bernadino, California
  - San Diego, California
  - San Fran Cisco, California
  - New Britain, Connecticut
  - New London, Connecticut
  - Leesburg, Florida
  - Miami, Florida
  - Miami Gardens, Florida
  - Pensacola, Florida
  - Tamarac, Florida
  - Tampa, Florida
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Naperville, Illinois
  - Springfield, Illinois
  - Wichita, Kansas
  - Witchita, Kansas
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Flowood, Mississippi
  - Kansas City, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Paramus, New Jersey
  - Willingboro, New Jersey
  - Buffalo, New York
  - New York, New York
  - Cleveland, Ohio
  - Middleburg Heights, Ohio
  - Willoughby, Ohio
  - Oklahoma City, Oklahoma
  - Allentown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - DeSoto, Texas
  - Irving, Texas
  - San Antonio, Texas
  - Wharton, Texas
  - Bothell, Washington
  - Spokane, Washington
- Rio Piedras, Puerto Rico

REFERENCES:
- [Derived] Lopena OJ, Alphs LD, Sajatovic M, Turkoz I, Sun L, Johnston KL, Sliwa JK, Najarian DM, Starr HL. Earlier Use of Long-Acting Injectable Paliperidone Palmitate Versus Oral Antipsychotics in Patients With Schizophrenia: An Integrated Patient-Level Post Hoc Analysis. J Clin Psychiatry. 2023 Sep 25;84(6):23m14788. doi: 10.4088/JCP.23m14788. PMID 37756123
- [Derived] Bell Lynum KS, Henderson DC, Wright HJ, Gogate JP, Kim E. Treatment Effect With Paliperidone Palmitate Compared With Oral Antipsychotics in Black/African American Patients With Schizophrenia and a History of Criminal Justice System Involvement: A Post Hoc Analysis of the PRIDE Study. J Clin Psychiatry. 2021 Feb 23;82(2):20m13356. doi: 10.4088/JCP.20m13356. PMID 33988924
- [Derived] Alphs L, Mao L, Lynn Starr H, Benson C. A pragmatic analysis comparing once-monthly paliperidone palmitate versus daily oral antipsychotic treatment in patients with schizophrenia. Schizophr Res. 2016 Feb;170(2-3):259-64. doi: 10.1016/j.schres.2015.12.012. Epub 2015 Dec 29. PMID 26742509
- [Derived] Alphs L, Bossie C, Mao L, Lee E, Starr HL. Treatment effect with paliperidone palmitate compared with oral antipsychotics in patients with recent-onset versus more chronic schizophrenia and a history of criminal justice system involvement. Early Interv Psychiatry. 2018 Feb;12(1):55-65. doi: 10.1111/eip.12271. Epub 2015 Sep 25. PMID 26403322
- [Derived] Alphs L, Benson C, Cheshire-Kinney K, Lindenmayer JP, Mao L, Rodriguez SC, Starr HL. Real-world outcomes of paliperidone palmitate compared to daily oral antipsychotic therapy in schizophrenia: a randomized, open-label, review board-blinded 15-month study. J Clin Psychiatry. 2015 May;76(5):554-61. doi: 10.4088/JCP.14m09584. PMID 25938474
- [Derived] Alphs L, Mao L, Rodriguez SC, Hulihan J, Starr HL. Design and rationale of the Paliperidone Palmitate Research in Demonstrating Effectiveness (PRIDE) study: a novel comparative trial of once-monthly paliperidone palmitate versus daily oral antipsychotic treatment for delaying time to treatment failure in persons with schizophrenia. J Clin Psychiatry. 2014 Dec;75(12):1388-93. doi: 10.4088/JCP.13m08965. PMID 25375367

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone Palmitate: Intramuscular injection, 234 milligram (mg) on Day 1, 156 mg on Day 8, followed by flexible monthly maintenance dosing as per investigator's discretion starting on Day 38 up to 15 months.
- Oral Antipsychotics: One of 7 oral antipsychotics (aripiprazole, haloperidol, olanzapine, paliperidone, perphenazine, quetiapine, and risperidone) that the investigator specified as appropriate for the participant was administered as per clinical practice for up to 15 months.
Period: Overall Study
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Started | 230 | 220
Treated | 226 | 218
Completed | 93 | 88
Not Completed | 137 | 132
Not completed — Adverse Event | 5 | 4
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 53 | 55
Not completed — Withdrawal by Subject | 37 | 27
Not completed — Physician Decision | 5 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Other | 32 | 36
Not completed — Noncompliance with Study Drug | 0 | 3
Not completed — Randomized but not Treated | 4 | 2

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) population included all participants who were randomly assigned to treatment and who received at least 1 dose of their randomly assigned study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics | Total
Number analyzed (Participants) | 226 | 218 | 444
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (10.57) | 38.6 (10.36) | 38.1 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 28 | 61
  Male | 193 | 190 | 383
Baseline Personal and Social Performance (PSP) Total Score [Mean (Standard Deviation); unit: Units on a scale] — The PSP score assesses degree of difficulty within 4 domains of behavior using 6-point Likert scale(0=absent to 5=very severe).The domain ratings were then transformed to PSP total score ranging from 1 to 100. Higher PSP total scores=better functioning.
  Units on a scale | 54.8 (12.83) | 55.0 (12.73) | 54.9 (12.76)
Baseline Clinical Global Impression - Severity (CGI-S) Total Score [Mean (Standard Deviation); unit: Units on a scale] — The CGI-S rating scale was a 7-point global assessment of symptom severity with scores determined by clinician as follows: 1=Not ill, 2=Very Mild, 3= Mild, 4= Moderate, 5= Marked, 6= Severe, and 7= Extremely Severe. The higher the score the worse the illness.
  Units on a scale | 3.8 (0.80) | 3.9 (0.70) | 3.8 (0.75)

OUTCOME MEASURES:

1. Primary Outcome: Time to First Treatment Failure
Description: Time to first treatment failure was the time from participant randomization to the first treatment failure, which was a composite endpoint consisting of any of the following events: arrest/incarceration, psychiatric hospitalization, discontinuation of antipsychotic treatment due to safety or tolerability, treatment supplementation with another antipsychotic due to inadequate efficacy, discontinuation of antipsychotic treatment due to inadequate efficacy, increase in level of psychiatric services to prevent imminent psychiatric hospitalization, suicide. A Treatment Failure Event Monitoring Board (EMB), blinded to individual participant treatment assignment, determined the occurrence and date of the first treatment failure event.
Time Frame: From date of randomization up to Month 15
Population: Explanatory Intent-to-Treat (eITT) population included all ITT participants who had their study assessments for time period between randomization date and eITT end point. The eITT end point for paliperidone palmitate was the last injection date+28 days and for oral antipsychotics was the last prescription date + the number of days' supply + 1 day.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 226 | 218
Days | 416 [285 to NA] — Upper limit of 95 percent (%) confidence interval was not estimable due to insufficient number of participants with event. | 226 [147 to 304]

2. Secondary Outcome: Time to First Psychiatric Hospitalization or Arrest/Incarceration
Description: A time to parameter looking only at 2 component events of treatment failure: arrest or incarceration, and psychiatric hospitalization. An arrest was defined as the taking of a participant into custody by legal authority, for any reason. Incarceration was defined as involuntary confinement by an officer of the law. Psychiatric hospitalization was an inpatient psychiatric hospitalization that occurred due to the participant's clinically significant worsening of symptoms of schizophrenia.
Time Frame: From date of randomization up to Month 15
Population: eITT population included all ITT participants who had their study assessments for time period between randomization date and eITT end point. The eITT end point for paliperidone palmitate was the last injection date+28 days and for oral antipsychotics was the last prescription date + the number of days' supply + 1 day.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 226 | 218
Days | NA [NA to NA] — Median and 95% confidence interval was not estimable due to insufficient number of participants with event. | 274 [202 to 407]

3. Secondary Outcome: Change From Baseline in Personal and Social Performance (PSP) Total Score During Overall Treatment Duration
Description: The PSP score assesses the degree of difficulty a participant exhibit over a 1 month period within 4 domains of behavior: a) socially useful activities, b) personal and social relationships, c) self-care, and d) disturbing and aggressive behavior. The investigators rate participants' degree of difficulty in each of the 4 domains using a 6-point Likert scale (from 0=absent to 5=very severe). The domain ratings were then transformed to PSP total score ranging from 1 to 100. Higher PSP total scores denote better functioning. A score between 71 and 100 represents normal to mild degree of dysfunction; a score between 31 and 70 represents varying degree of difficulty; and a score <=30 represents poor function that requires intensive supervision.
Time Frame: Baseline up to Month 15
Population: eITT population. 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 203 | 185
Units on a scale | 5.75 (0.690) | 5.36 (0.690)

4. Secondary Outcome: Time to First Psychiatric Hospitalization
Description: A time-to parameter looking only at 1 component event of treatment failure: psychiatric hospitalization. Time to first psychiatric hospitalization was admission date of the psychiatric hospitalization recorded in the "Assessment of Treatment Failure - Psychiatric Hospitalization."
Time Frame: From date of randomization up to Month 15
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 226 | 218
Days | NA [NA to NA] — Median and 95% confidence interval was not estimable due to insufficient number of participants with event. | NA [NA to NA] — Median and 95% confidence interval was not estimable due to insufficient number of participants with event.

5. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score During Overall Treatment Duration
Description: The CGI-S rating scale was a 7-point global assessment of symptom severity with scores determined by clinician as follows: 1=Not ill, 2=Very Mild, 3= Mild, 4= Moderate, 5= Marked, 6= Severe, and 7= Extremely Severe. The higher the score the worse the illness.
Time Frame: Baseline up to Month 15
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 219 | 205
Units on a scale | -0.48 (0.038) | -0.43 (0.037)

6. Primary Outcome: Percentage of Participants in Each Event Category of First Treatment Failure
Description: First treatment failure was a composite endpoint consisting of any of the following events: arrest/incarceration, psychiatric hospitalization, discontinuation (D/C) of antipsychotic treatment due to safety or tolerability, treatment supplementation with another antipsychotic due to inadequate efficacy, discontinuation of antipsychotic treatment due to inadequate efficacy, increase in level of psychiatric services to prevent imminent psychiatric hospitalization, suicide. A Treatment Failure Event Monitoring Board (EMB), blinded to individual participant treatment assignment, determined the occurrence and date of the first treatment failure event. Percentage of participants who experienced treatment failure due to any event and for each specific category of event were assessed.
Time Frame: From date of randomization up to Month 15
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Number analyzed (Participants) | 226 | 218
percentage of participants
  Treatment Failure Due to Any Event | 39.8 | 53.7
  Arrest/incarceration | 21.2 | 29.4
  Psychiatric hospitalization | 8.0 | 11.9
  D/C due to safety/tolerability | 6.6 | 3.7
  Treatment supplementation | 2.2 | 2.8
  D/C due to inadequate efficacy | 0.4 | 4.1
  Increase in level of psychiatric services | 1.3 | 1.8
  Suicide | 0 | 0

ADVERSE EVENTS:
Description: Intent to Treat (ITT) population included all participants who were randomly assigned to treatment and who received at least 1 dose of their randomly assigned study treatment.
Arm/Group | Paliperidone Palmitate | Oral Antipsychotics
Serious Adverse Events (participants affected / at risk) | 42/226 | 53/218
Other Adverse Events (participants affected / at risk) | 178/226 | 155/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Palmitate (N=226) | Oral Antipsychotics (N=218)
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Drug Withdrawal Syndrome (General disorders) | 0 | 1
Non-cardiac Chest Pain (General disorders) | 1 | 0
Sudden Death (General disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Acquired Immunodeficiency Syndrome (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1
Cholecystitis Infective (Infections and infestations) | 0 | 1
H1N1 Influenza (Infections and infestations) | 1 | 0
HIV Infection (Infections and infestations) | 1 | 0
Otitis Media (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Wound Infection (Infections and infestations) | 0 | 1
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Gun Shot Wound (Injury, poisoning and procedural complications) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Intentional Overdose (Injury, poisoning and procedural complications) | 1 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Perirenal Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 1 | 0
Traumatic Lung Injury (Injury, poisoning and procedural complications) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastric Cancer Stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Akathisia (Nervous system disorders) | 1 | 0
Cerebellar Ataxia (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Dystonia (Nervous system disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Facial Paresis (Nervous system disorders) | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Acute Psychosis (Psychiatric disorders) | 1 | 2
Aggression (Psychiatric disorders) | 0 | 1
Agitation (Psychiatric disorders) | 2 | 0
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 2 | 1
Alcoholism (Psychiatric disorders) | 2 | 0
Delusion (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 4 | 1
Depression Suicidal (Psychiatric disorders) | 1 | 0
Depressive Symptom (Psychiatric disorders) | 1 | 0
Factitious Disorder (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Hallucination, Auditory (Psychiatric disorders) | 1 | 1
Hallucinations, Mixed (Psychiatric disorders) | 1 | 0
Homicidal Ideation (Psychiatric disorders) | 0 | 3
Mania (Psychiatric disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 2 | 0
Polysubstance Dependence (Psychiatric disorders) | 0 | 1
Psychotic Behaviour (Psychiatric disorders) | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 11 | 7
Schizoaffective Disorder Bipolar Type (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 4 | 11
Schizophrenia, Paranoid Type (Psychiatric disorders) | 4 | 5
Substance Abuse (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 5 | 11
Suicide Attempt (Psychiatric disorders) | 1 | 3
Renal Failure Acute (Renal and urinary disorders) | 1 | 2
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Status Asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Palmitate (N=226) | Oral Antipsychotics (N=218)
Hyperprolactinaemia (Endocrine disorders) | 7 | 4
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 5
Constipation (Gastrointestinal disorders) | 7 | 8
Diarrhoea (Gastrointestinal disorders) | 4 | 7
Dry Mouth (Gastrointestinal disorders) | 15 | 18
Dyspepsia (Gastrointestinal disorders) | 7 | 3
Nausea (Gastrointestinal disorders) | 9 | 6
Salivary Hypersecretion (Gastrointestinal disorders) | 7 | 0
Toothache (Gastrointestinal disorders) | 11 | 13
Vomiting (Gastrointestinal disorders) | 2 | 5
Fatigue (General disorders) | 17 | 6
Injection Site Pain (General disorders) | 42 | 0
Irritability (General disorders) | 4 | 6
Pain (General disorders) | 1 | 5
Bronchitis (Infections and infestations) | 6 | 5
Influenza (Infections and infestations) | 4 | 5
Nasopharyngitis (Infections and infestations) | 15 | 14
Upper Respiratory Tract Infection (Infections and infestations) | 13 | 11
Joint Sprain (Injury, poisoning and procedural complications) | 2 | 6
Laceration (Injury, poisoning and procedural complications) | 4 | 12
Blood Prolactin Increased (Investigations) | 11 | 2
Semen Volume Decreased (Investigations) | 5 | 0
Weight Increased (Investigations) | 30 | 16
Abnormal Weight Gain (Metabolism and nutrition disorders) | 11 | 4
Increased Appetite (Metabolism and nutrition disorders) | 16 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 13 | 8
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 5 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 9 | 8
Akathisia (Nervous system disorders) | 26 | 17
Dizziness (Nervous system disorders) | 6 | 11
Dyskinesia (Nervous system disorders) | 6 | 4
Dystonia (Nervous system disorders) | 5 | 5
Extrapyramidal Disorder (Nervous system disorders) | 5 | 4
Headache (Nervous system disorders) | 17 | 19
Sedation (Nervous system disorders) | 15 | 18
Somnolence (Nervous system disorders) | 10 | 16
Tremor (Nervous system disorders) | 5 | 3
Agitation (Psychiatric disorders) | 5 | 5
Anxiety (Psychiatric disorders) | 25 | 18
Depression (Psychiatric disorders) | 19 | 17
Hallucination, Auditory (Psychiatric disorders) | 3 | 6
Insomnia (Psychiatric disorders) | 42 | 27
Libido Decreased (Psychiatric disorders) | 13 | 3
Schizophrenia (Psychiatric disorders) | 7 | 6
Suicidal Ideation (Psychiatric disorders) | 4 | 9
Amenorrhoea (Reproductive system and breast disorders) | 5 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 17 | 1
Galactorrhoea (Reproductive system and breast disorders) | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Hypertension (Vascular disorders) | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days